CLINICAL TRIAL: NCT02098460
Title: To Compare the Effect of Concomitant Administration of Probucol and Cilostazol With Probucol Single Treatment on the Atherosclerosis Related Markers (Including the Thickness of the Achilles Tendon) and Evaluate Safety (Based on Atorvastatin Treatment) in Severe Hypercholesterolemia Subject
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 260-13-806-01
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2014-03

CONDITIONS: Severe Hypercholesterolemia
Keywords: the Achilles tendon; intima-media thickness
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Probucol; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probucol,Cilostazol (Placebo Comparator): Atorvastatin + Probucol-placebo + Cilostazol-placebo
  Interventions: Drug: Atorvastatin, Probucol, Cilostazol
- Cilostazol (Placebo Comparator): Atorvastatin + Probucol+ Cilostazol-placebo
  Interventions: Drug: Atorvastatin, Probucol, Cilostazol
- Probucol, Cilostazol (Active Comparator): Atorvastatin + Probucol + Cilostazol
  Interventions: Drug: Atorvastatin, Probucol, Cilostazol

INTERVENTIONS:
Drug: Atorvastatin, Probucol, Cilostazol

SUMMARY:
To evaluate the effect of concomitant administration of Probucol and Cilostazol (based on Atorvastatin treatment) on the atherosclerosis related markers (including the thickness of the Achilles tendon) in severe hypercholesterolemia subject, through the observation of the thickness of the Achilles tendon, the thickness of mean carotid intima-media, anti-oxidation biomarkers and serum lipid profile.

DETAILED DESCRIPTION:
Multicenter, randomized, controlled, single-blinded, three parallel arms study. Group A: Atorvastatin + Probucol-placebo + Cilostazol-placebo Group B: Atorvastatin + Probucol + Cilostazol-placebo Group C: Atorvastatin + Probucol + Cilostazol

ELIGIBILITY:
Inclusion Criteria:

1. The subject whose voluntary written informed consent is obtained for participation in this study;
2. 18≤age≤70；
3. The subject with low-density lipoprotein cholesterol (LDL-C) ≥ 4.66 mmol/L (180 mg/dL) (the highest level either pre-treatment or on treatment);
4. The subject with ATT≥9mm.

Exclusion Criteria:

1. The subject with homozygous familial hyperlipidemia;
2. The subject who took Probucol within 6 months before the screening test;
3. The subject who took Cilostazol within 1 month before the screening test;
4. The subject who took Ezetimibe within 1 month before the screening test;
5. The subject who hoped to treat with Ezetimibe within this study period;
6. The subject being treated with Cyclosporine;
7. The subject with a history of hypersensitivity to Probucol and Cilostazol;
8. The subject with a triglyceride (TG) level greater than 4.52 mmol/L (400 mg/dL);
9. The subject with diabetes: HbA1c level greater than 8.4% (NGSP);
10. The subject with New York Heart Association (NYHA) classification: Class III and IV;
11. The subject with a QTc interval greater than 450 msec (male) or 470 msec (female);
12. The subject with serious ventricular arrythmias (frequent episodes of multifocal ventricular extrasystole);
13. The subject with atrial fibrillation (including paroxysmal atrial fibrillation);
14. The subject with congestive cardiac failure or unstable angina;
15. The subject with liver and renal functions that satisfy the following criteria within 28 days prior to start of the investigational medicinal product (IMP) administration.

    * AST ≥100 IU/L, ALT≥100 IU/L
    * Serum creatinine ≥1.5 mg/dL (133 µmol/L)
16. The subject who are participating in another clinical trial;
17. Woman during pregnancy or potential pregnancy, and breastfeeding;
18. Women of childbearing potential who are not agree to use an appropriate method of contraception;
19. The subject who are not considered by the Investigators to be appropriate to participate in this study for any other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
the effect of concomitant administration of Probucol and Cilostazol on the mean achilles tendon thickness (ATT) | at Month 6, 12 and 24

SECONDARY OUTCOMES:
the additional effect of concomitant administration of Probucol and Cilostazol on mean carotid intima-media thickness (IMT) | at Month 12 and 24
the preventive effect of concomitant administration of Probucol and Cilostazol on the incidence of cerebrovascular and cardiovascular events (including intervention) | 2 years
the effect of concomitant administration of Probucol and Cilostazol on biomarkers | 2 years
the safety of Probucol or concomitant administration of Probucol and Cilostazol as determined by physical examination, vital signs, adverse events (AEs), laboratory examinations and 12-lead electrocardiogram (ECGs) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Lin, Dr, Principal Investigator — Anzhen hospital
Locations (1):
- Anzhen hospital, Beijing, China